CLINICAL TRIAL: NCT03126864
Title: A Phase 1 Safety Study of Adoptive Cellular Therapy Using Autologous T Cells Transduced With Lentivirus to Express a CD33 Specific Chimeric Antigen Receptor in Patients With Relapsed or Refractory CD33-Positive Acute Myeloid Leukemia
Brief Title: Study of Adoptive Cellular Therapy Using Autologous T Cells Transduced With Lentivirus to Express a CD33 Specific Chimeric Antigen Receptor in Patients With Relapsed or Refractory CD33-Positive Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated per the PI's request.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Intrexon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0341; NCI-2018-01167 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Hematopoietic/Lymphoid Cancer; Acute Myeloid Leukemia
Keywords: Hematopoietic/Lymphoid Cancer; Acute Myeloid Leukemia; AML; Relapsed or Refractory CD33-Positive; CD33-CAR-T cells; Fludarabine; Fludarabine phosphate; Fludara; Cyclophosphamide; Cytoxan; Neosar
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Recurrence | interventions — Leukapheresis; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CD33-CAR-T cells - Adult Group (Experimental): After enrollment, steady state leukapheresis performed to collect apheresis material.
  Fludarabine administered by vein on Days -5 to -3.
  Cyclophosphamide administered by vein on Day -3.
  CD33-CAR-T cell infusion administered by vein on Day 0. First group of participants receive the lowest dose level. Each new group will receive a higher dose than the one before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of T-cells is found.
  Interventions: Procedure: Leukapheresis; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CD33-CAR-T Cell Infusion
- CD33-CAR-T cells - Pediatric Group (Experimental): After enrollment, steady state leukapheresis performed to collect apheresis material.
  Fludarabine administered by vein on Days -5 to -3.
  Cyclophosphamide administered by vein on Day -3.
  CD33-CAR-T cell infusion administered by vein on Day 0. First group of participants receive the lowest dose level. Each new group will receive a higher dose than the one before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of T-cells is found.
  Interventions: Procedure: Leukapheresis; Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CD33-CAR-T Cell Infusion

INTERVENTIONS:
Procedure: Leukapheresis — After enrollment, steady state leukapheresis performed to collect apheresis material. The goal is to achieve a target total nucleated cell (TNC) yield of at least 5 x 10^9 (expected range 5 x 10^8 - 5 x 10^10), for up to two days.
Drug: Fludarabine — 25 mg/m2 administered by vein on Days -5 to -3.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Cyclophosphamide — 900 mg/m2 administered by vein on Day -3.
  Other Names: Cytoxan; Neosar
Biological: CD33-CAR-T Cell Infusion — CD33-CAR-T cell infusion administered by vein on Day 0. First group of participants receive the lowest dose level. Each new group will receive a higher dose than the one before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of T-cells is found. Starting dose level is > 1.5 x 105/kg but ≤ 4.5 x 105/kg.

SUMMARY:
Any time the words "you," "your," "I," or "me" appear, it is meant to apply to the potential participant.

The goal of this clinical research study is to learn about the safety and tolerability of 3 different doses of CD33-CAR-T cells (referred to throughout the consent as "T-cells") in patients who have CD33-positive acute myeloid leukemia (AML) that is relapsed (has come back) or refractory (has not responded to treatment).

CD33-CAR-T is made by genetically modifying (changing) your T-cells (a type of white blood cell). T-cells are genetically changed to help target leukemia cells.

This is an investigational study. CD33-CAR-T is not FDA approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how the study drug is designed to work.

Up to 39 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1-80 years of age. The pediatric cohort is defined as age younger than 18 years.
2. Patients with active (blood or bone marrow blasts >5%) relapsed or refractory CD33+ acute myeloid leukemia (AML) de novo, or secondary. a. Relapsed AML is defined as patients that had a first complete remission (CR) before developing recurrent disease. b. Refractory AML defined as patients that have not achieved a CR after 2 cycles of induction chemotherapy.
3. Patients must have bone marrow and peripheral blood studies available for confirmation of diagnosis of AML; CD33 positivity must be confirmed by either flow cytometry or immunohistochemistry; cytogenetics, flow cytometry, and molecular studies (such as FMS-like tyrosine kinase-3 [Flt-3] status) will be obtained as per standard practice.
4. ECOG performance status score </= 2.
5. Pretreatment calculated or measured creatinine clearance (absolute value) of >= 60 mL/minute.
6. Serum bilirubin =< 3.0 mg/dL.
7. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 5 times the institutional upper limits of normal.
8. Ejection fraction measured by echocardiogram (ECHO) or multi gated acquisition scan (MUGA) >50%.
9. Subject does not require supplemental oxygen or mechanical ventilation, and oxygen saturation by pulse oximetry is 94% or higher on room air.
10. Negative serum pregnancy test.
11. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately.
12. Patients who have undergone allo-SCT are eligible if they are at least 3 months post SCT, have relapsed AML, are not on treatment or prophylaxis for GVHD, and have no active GVHD.
13. All patients or legally responsible parent or guardian must have the ability to understand and willingness to sign a written informed consent

Exclusion Criteria:

1. Diagnosis of acute promyelocytic leukemia (APL M3): t(15;17)(q22;q12); (promyelocytic leukemia [PML]/retinoic acid receptor [RAR] alpha [a]) and variants excluded.
2. Patients with extramedullary disease as their sole site of relapsed AML.
3. Acceptable allogeneic stem cell donor with imminent plans to proceed with allo-SCT.
4. Known central nervous system (CNS) leukemic involvement that is refractory to intrathecal chemotherapy and/or cranio-spinal radiation; patients with a history of CNS disease that have been effectively treated to complete remission (< 5 white blood cell [WBC]/mm^3 and no blasts in cerebrospinal fluid [CSF]) will be eligible.
5. Ongoing or active or uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, poorly controlled pulmonary disease or psychiatric illness/social situations that would limit compliance with study requirements.
6. Human immunodeficiency virus (HIV) seropositivity, or active hepatitis B or C infection based on testing performed within 4 weeks of enrollment.
7. Currently enrolled in another investigational therapy protocol for AML.
8. Participants with presence of other active malignancy within 2 years of study entry; participants with history of prior malignancy treated with curative intent and achieved CR within 2 years are eligible.
9. Pregnant and lactating women are excluded from this study
10. Failure of research participant or legally responsible parent or guardian to understand the basic elements of the protocol and/or the risks/benefits of participating in this phase I study.
11. History of allergic reactions attributed to compounds of similar chemical or biological composition to cetuximab (anti-EGFR).
12. History of allergic reactions to products containing mouse and bovine protein antibodies.
13. Receiving corticosteroids at >20 mg (age >17) or >0.5mg/kg (age <18) daily prednisone dose or equivalent.
14. Active autoimmune disease requiring systemic immunosuppressive therapy.
15. Patient, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Recommended Phase II Dose (RP2D) of CD33-CAR-T Cells | 28 days after completion of the CD33-CAR-T infusion
  RP2D defined as the highest dose level in which 6 patients have been treated with at most 1 instance of dose limiting toxicity (DLT).
  DLT is defined as a clinically significant adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications and occurring during the first course on study that meets any of the following criteria:
  * CTCAE grades non-reversible grade 3, or any grade 4-5 allergic reactions related to the study cell infusion.
  * CTCAE grades non-reversible grade 3, or any grade 4-5 autoimmune reactions related to the study cell infusion.
  * CTCAE grades non-reversible grade 3, or any grade 4-5 organ toxicity (cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary, or neurologic) not pre-existing or due to the underlying malignancy and occurring within 28 days of study product infusion related to study cell infusion.

SECONDARY OUTCOMES:
Disease Response to CD33-CAR-T Cells | On Day 7, at Weeks 2, 4, and 8, and at Months 3, 6, and 12 after CD33-CAR-T Cell infusion
  Response to treatment evaluated according to the World Health Organization (WHO) standardized response criteria for myelodysplastic syndromes.
  Disease response to CD33-CAR-T cells defined as Complete Remission (CR), Complete Remission without Platelet Recovery (CRp), Complete Remission without Neutrophil Recovery (CRn), Complete Remission with Incomplete Blood Count Recovery (CRi), Partial Remission (PR) or Non-responder (NR).

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, MD, PHD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org